CLINICAL TRIAL: NCT06810401
Title: Impact of Smoking on Macrophage-Related Chemokines During Initial Peri-implantitis
Brief Title: Effect of Smoking on Macrophage-related Chemokines Before and After Non-surgical Treatment of Initial Peri-implantitis
Acronym: PICF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buse Naz BÜYÜKAKÇALI ALTAY (Other)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor-Investigator, Buse Naz BÜYÜKAKÇALI ALTAY, Principal Investigator, Research Assistant, Gazi University
Organization: Gazi University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-KD24/01
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Peri-implantitis
Keywords: Peri-implantitis; Smoking; Chemokines
MeSH Terms: conditions — Peri-Implantitis; Smoking | interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peri-implantitis patients (Experimental): All peri-implantitis patients in both smoking and non-smoking groups received full-mouth non-surgical periodontal treatment using sterile ultrasonic scalers (Woodpecker Piezo Cavitron Ultrasonic Scaler Handpiece (HW-5L), EMS, Switzerland)), currets (Lsh6-h7, Osung MND, Korea), and sterile saline irrigations. Non-surgical treatment of peri-implantitis involves the debridement of hard- and soft accumulations on implant surfaces using titanium curettes (Titanium Implant Scaler 204SD, Hu-Friedy) for 15 minutes, followed by irrigation with sterile saline solution
  Interventions: Procedure: Debridement of implant surface with titanium curettes and irrigation with sterile saline solution

INTERVENTIONS:
Procedure: Debridement of implant surface with titanium curettes and irrigation with sterile saline solution — All patients in both groups received non-surgical treatment of peri-implantitis involving the debridement of hard- and soft accumulations on implant surfaces using titanium curettes (Titanium Implant Scaler 204SD, Hu-Friedy) for 15 minutes, followed by irrigation with sterile saline solution
  Other Names: Non-surgical treatment of peri-implantitis

SUMMARY:
Peri-implantitis is a condition affecting tissues around dental implants, leading to inflammation and bone loss. Smoking is a known risk factor that increases the risk of developing peri-implantitis and reduces treatment success. Smokers often have worse outcomes after treatment compared to non-smokers.

Macrophage activity is crucial for fighting infections, but smoking can impair their function, leading to tissue damage. Smoking reduces blood flow and oxygen levels in tissues, hindering healing. Specific chemokines (CCL-2, CCL-8, CXCL-9, and CCL-3) help direct immune responses by recruiting macrophages and other immune cells to infection sites. Understanding how smoking affects these chemokines is essential for improving peri-implantitis treatment outcomes. Peri-implantitis is a complex condition caused by various factors, which makes it challenging to study how smoking affects the immune response in advanced stages of the disease. This study aims to investigate how smoking influences specific chemical signals associated with the immune response (CCL-2, CCL-8, CCL-3, and CXCL-9) in the fluid around dental implants, both before and after non-surgical treatment. The research will compare smokers to non-smokers during the early stages of peri-implantitis.

DETAILED DESCRIPTION:
1. Ethics Approval and Determination of Sample Size

   The study was approved by the Clinical Research Ethics Committee of Başkent University, Ankara, Türkiye (Study protocol number: D-KD24/01) in accordance with the Helsinki Declaration of 1975, as revised in 2013.

   The power analysis was conducted using GPower software. Based on previous research comparing pre- and post-treatment MIP-1α levels in PICF samples, the required minimum sample size was calculated to be 52 participants, with 26 participants in each group in order to achieve a power of 80% (effect size f = 0.2; α error = 0.05). Estimating a drop-out rate of 20%, the present study aimed to recruit 63 patients.
2. Study Design

   Study planning, patient recruitment, treatments, and sample collection were performed at the clinics of the Department of Periodontology, Faculty of Dentistry, Gazi University, Türkiye, between January 2024 and October 2024. All individuals who were diagnosed with peri-implantitis (peri-implant bleeding on probing (BOP+) and/or suppuration, PPD of ≥ 6 mm, and radiographic crestal bone loss of ≥ 3 mm apical of the most coronal portion of the intraosseous part of the dental implant at their initial visit at the periodontology clinics of Gazi University Faculty of Dentistry, were invited to take part in the study.
3. Inclusion and Exclusion Criteria

   Inclusion criteria were: 1) willingness to participate in the study, 2) having a dental implant that was loaded at least one year before the initiation of the study, that was diagnosed with peri-implantitis, and that has PD of 6-7 mm, 3) the implants had been in function for at least 1 years. Exclusion criteria were: 1) having received periodontal therapy or any oral decontamination treatment or received antibiotics or steroids in the last six months before the initiation of the study, 2) being pregnant or breastfeeding, 3) being diagnosed with rheumatoid arthritis, lupus erythematosus, poorly controlled systemic diseases (such as diabetes or hypertension), 4) having a medical history of radiation or cancer therapy.
4. Study population

   Comprehensive periodontal and radiographic examinations of the teeth and dental implants were performed for all participants at baseline. Site-level clinical parameters were measured at four sites of each implant (mesial, buccal, distal, and lingual/palatal). The measurements included PPD (mm), BOP, visible plaque index (VPI), and width of peri-implant keratinized tissue (≥ 2 mm or < 2 mm) assessments. Peri-apical radiographs were obtained to measure peri-implant radiographic bone level. All clinical measurements were performed using a periodontal probe. All measurements were conducted by the same investigator. Patients who had PPD ≥ 8 mm around their implants were excluded from the study.

   A total of 63 peri-implantitis patients who met the inclusion and exclusion criteria were recruited for the study. All participants were provided verbal and written information regarding the nature of the study, and written informed consent was obtained from each participant. The study population was later divided into two groups based on self-reported cigarette smoking. Smokers were individuals who reported smoking at least one cigarette per day for at least one year (smoking peri-implantitis patients (SPI), n = 30), while never-smokers were individuals who had never used tobacco in any form (non-smoking peri-implantitis patients (NSPI), n = 33).
5. Peri-implant and Periodontal Treatment

   All patients in both groups received full-mouth non-surgical periodontal treatment using sterile ultrasonic scalers (Woodpecker Piezo Cavitron Ultrasonic Scaler Handpiece (HW-5L), EMS, Switzerland)), currets (Lsh6-h7, Osung MND, Korea), and sterile saline irrigations. Non-surgical treatment of peri-implantitis involved the debridement of hard- and soft accumulations on implant surfaces using titanium curettes (Titanium Implant Scaler 204SD, Hu-Friedy) for 15 minutes, followed by irrigation with sterile saline solution. Infiltration anesthesia was used if requested by the patient. Customized oral hygiene instructions were given to all participants after treatment. After 2 months (8 weeks), patients received a call for a control visit, including a supragingival debridement and oral hygiene instructions. All clinical and radiographic measurements were repeated 4 months after the completion of their non-surgical peri-implant treatment.
6. Sample Collection PICF samples were collected from all participants before (T0) and 4 months after (T1) peri-implant non-surgical treatment. A 30-second sampling protocol was used. Before sampling, the sample area was isolated with cotton rolls and dried using a gentle stream of air. A single PICF sample was collected from each implant pocket using PerioPaper strips (Oralflow Inc., New York, USA). These paper strips were placed 1-2 mm under the crevice of the pocket and kept for precisely 30 seconds. To minimize evaporation, volume quantification was performed immediately after sampling using a Periotron 8000 device (Oralflow Inc., New York, USA). The Periotron 8000 was calibrated before starting the study and recalibrated periodically. After quantifying the PICF volume, each paper strip was placed in a dry Eppendorf tube. The samples were stored at -80°C until being transferred in dry ice to the University of Turku, Institute of Dentistry, Finland, for biochemical analyses.
7. Biomarker Analysis

Each PICF sample was eluted in 200 µl of phosphate-buffered saline (PBS) containing 0.5% bovine serum albumin. The tubes were then centrifuged at 10,000 g at 4°C for 10 minutes. The CCL-2, CCL-8, CCL-3, and CXCL-9 concentrations were detected with Luminex® 200™ using multiplex immunoassay kits (Bio-Plex Pro™ Human Chemokine Assays, Bio-Rad Laboratories, California, USA) according to the manufacturer's recommendations. Concentrations (pg/ml) were converted to the mediator amount collected at 30 seconds (pg/30 s). The lower limits of quantification (LLOQ) for each chemokine were as follows: 0.3 pg/ml for CCL-2, 0.03 pg/ml for CCL-8, 0.4 pg/ml for CCL-3, and 1.8 pg/ml for CXCL-9.

8. Statistical Analysis

Data analysis was performed using IBM SPSS Statistics (Version 29.0 for Windows; IBM Corp). The normality of the outcomes was evaluated with the Shapiro-Wilk test. Group differences in categorical variables were assessed using the Pearson Chi-square test, while age distribution between groups was compared using the Independent Samples t-test. The Mann-Whitney U test was applied to compare clinical and biochemical outcomes between groups. To compare baseline (T0) and 4-month post-operative (T1) outcomes of biochemical and clinical variables within each group, the Wilcoxon signed-rank test was used. Repeated measures analysis of variance test (controlled for age) was used to determine whether there is a difference in the effectiveness of treatment over time. Logarithmic conversions (Log10) were applied to chemokine levels (pg/30 s) before the repeated measures analysis of the variance test. A p-value of < 0.05 was considered to be statistically significant for all the parameters. A four-parameter logistic regression model was used to calculate chemokine concentrations in PICF. CCL-2 was detected in all samples, while CCL-8 was below the limit of detection (LOD) in 77 samples (T0: 55%, T1: 85%), CCL-3 in 30 samples (T0: 15%, T1: 40%), and CXCL-9 in 26 samples (T0: 15%, T1: 34%). In descriptive analyses, due to a high number of missing data, CCL-8 was excluded from statistical comparisons, while CCL-3 and CXCL-9 concentrations below the regression curve were substituted with a value equal to half of their lowest limit of quantification (LOD/2)

ELIGIBILITY:
Inclusion Criteria:

1. willingness to participate in the study
2. having a dental implant that was loaded at least one year before the initiation of the study, that was diagnosed with peri-implantitis, and that has PD of 6-7 mm, 3) the implants had been in function for at least 1 year.

Exclusion Criteria:

1. having received periodontal therapy or any oral decontamination treatment or received antibiotics or steroids in the last six months before the initiation of the study,
2. being pregnant or breastfeeding,
3. being diagnosed with rheumatoid arthritis, lupus erythematosus, poorly controlled systemic diseases (such as diabetes or hypertension),
4. having a medical history of radiation or cancer therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Biochemical Outcomes | Assessment and comparison of peri-implant crevicular fluid chemokine levels before and four months after non-surgical treatment of initial peri-implantitis in smoking and non-smoking individuals
  Analysis and comparison of peri-implant crevicular fluid levels of CCL-2, CCL-3, and CXCL-9 before and after non-surgical treatment of initial peri-implantitis in smokers and non-smokers.

SECONDARY OUTCOMES:
Probing Pocket Depth (mm) | Assessment and comparison of clinical outcomes for non-surgical treatment of peri-implantitis before and after four months.
  Assessment: Probing pocket depth was measured using a periodontal probe Unit of Measure: Millimeters (mm). Criteria: A reduction in probing pocket depth to 5 mm or less after four months indicates a healthy outcome.
Bleeding on Probing | Assessment and comparison of clinical outcomes for non-surgical treatment of peri-implantitis before and after four months.
  Assessment: The presence of bleeding during probing was evaluated with a periodontal probe Unit of Measure: The bleeding status was categorized as 1 = bleeding on probing and 0 = absence of bleeding.
  Criteria: The presence of bleeding in the pocket area is viewed as an unsatisfactory healing outcome.
Visible Plaque Score | Assessment and comparison of clinical outcomes for non-surgical treatment of peri-implantitis before and after four months.
  Assessment: The presence of visible plaque was evaluated with a periodontal probe Unit of Measure: The presence of plaque was categorized as 1= presence of plaque and 0= absence of plaque.
  Criteria: The presence of plaque indicates an unsatisfactory healing outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ulvi K GURSOY, Prof., Study Director — University of Turku
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altay BNB, Cankaya ZT, Yilmaz M, Gursoy M, Bodur A, Gursoy UK. Impact of Smoking on Macrophage-Related Chemokines During Initial Peri-Implantitis: A Prospective Cohort Study. Clin Implant Dent Relat Res. 2025 Jun;27(3):e70052. doi: 10.1111/cid.70052. PMID 40399133